CLINICAL TRIAL: NCT00725933
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of BIIB028 Administered to Subjects With Advanced Solid Tumors
Brief Title: Administration of BIIB028 to Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121ST101
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — HSP90 Heat-Shock Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BIIB028 — IV infusion administered twice weekly until disease progression or unacceptable toxicity

SUMMARY:
Safety and Tolerability of BIIB028

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Age greater than or equal to 18 years at the time of informed consent.
* Subjects with histological or cytological confirmed solid tumors who have failed standard therapies or for which no standard therapy is available.
* Anticipated survival of at least 3 months in the opinion of the Investigator.
* ECOG performance status of less than or equal to 2.
* Lab values consistent with adequate renal hepatic and bone marrow function.
* Must utilize effective contraception.

Exclusion Criteria:

* Pregnant (positive pregnancy test) or nursing women
* Prior treatment with Hsp90 inhibitors at any time.
* Prior antitumor therapies including prior experimental agents, approved antitumor small molecules and biologics, or radiotherapy with in 28 days or <3 half lives (whichever is longer). In addition,prior to enrollment, all asociated toxicities must have been resolved to eligibility levels.
* Concurrent severe or uncontrolled other medical disease (i.e, diabetes, hypertension, coronary artery disease, congestive heart failure), which in the opinion of the Investigator and/ or the Sponsor could compromise assessment of safety.
* Use of anticoagulants, except low dose warfarin.
* History of seizure, previous significant head trauma (e.g., associated with loss of consciousness for more than 5 minutes), abrupt discontinuation of benzodiazepines, or use of potentially epileptogenic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of BIIB028 | As specified in Protocol

SECONDARY OUTCOMES:
PK and PD of BIIB028 | As specified in protocol
Antitumor activity | As specified in protocol

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Encinitas, California
  - Research Site, Los Angeles, California
  - Research Site, Houston, Texas

REFERENCES:
- [Background] Hong D, Said R, Falchook G, Naing A, Moulder S, Tsimberidou AM, Galluppi G, Dakappagari N, Storgard C, Kurzrock R, Rosen LS. Phase I study of BIIB028, a selective heat shock protein 90 inhibitor, in patients with refractory metastatic or locally advanced solid tumors. Clin Cancer Res. 2013 Sep 1;19(17):4824-31. doi: 10.1158/1078-0432.CCR-13-0477. Epub 2013 Jul 19. PMID 23873691